CLINICAL TRIAL: NCT02401399
Title: Preoperative Regular Diet of 900 Kcal/Day vs Balanced Energy High Protein Formula vs Immunonutrition Formula: Effect on Postoperative Pain After Laparoscopic Sleeve Gastrectomy
Brief Title: Preoperative Diet Before Sleeve Gastrectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, MD, PhD, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HGUE15-2
Record Dates: First submitted 2015-03-24; First posted 2015-03-27 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Diet; Immunonutrition Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- regular diet (Placebo Comparator): The patients receive regular diet of 900 Kcal/day during 15 days before surgery
  Interventions: Dietary Supplement: Regular diet
- high protein formula (Active Comparator): The patients receive high protein formula during 15 days before surgery
  Interventions: Dietary Supplement: High protein formula
- Immunonutrition (Experimental): The patients receive Immunonutrition during 15 days before surgery
  Interventions: Dietary Supplement: Immunonutrition

INTERVENTIONS:
Dietary Supplement: Regular diet — The patients receive regular diet 900 Kcal/day during 15 days before surgery
  Arms: regular diet
Dietary Supplement: High protein formula — The patients receive high protein formula during 15 days before surgery
  Arms: high protein formula
Dietary Supplement: Immunonutrition — The patients receive Immunonutrition formula during 15 days before surgery
  Arms: Immunonutrition

SUMMARY:
Patients undergoing sleeve gastrectomy aara randomized into 3 groups:preoperative regular diet , preoperative balanced energy high protein formula and Immunonutrition formula.Postoperative pain and acute phase reactants at 24hours after surgery are investigated.

DETAILED DESCRIPTION:
Patients undergoing sleeve gastrectomy as bariatric procedure ara randomized into 3 groups: those patients receiving a preoperative regular diet of 900 Kcal/day (Group 1), those receiving preoperative balanced energy high protein formula (Group 2) and those receiving preoperative Immunonutrition formula (Group 3). Postoperative pain and acute phase reactants at 24hours after surgery are investigated.

ELIGIBILITY:
Inclusion Criteria:

* BMI >40 Kg/m2
* BMI > 35 Kg/m2 with the presence of comorbidities associated to obesity

Exclusion Criteria:

* gastroesophageal reflux
* patients with uncontrolled psychiatric disorders
* active infections or malignancies
* other concomitant pathology considered as a contraindication for bariatric surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 24 hours after surgery

SECONDARY OUTCOMES:
C reactive protein | 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Ruiz Tovar, Principal Investigator — Hospital General Elche

REFERENCES:
- [Derived] Ruiz-Tovar J, Zubiaga L, Diez M, Murcia A, Boix E, Munoz JL, Llavero C; OBELCHE group. Preoperative Regular Diet of 900 kcal/day vs Balanced Energy High-Protein Formula vs Immunonutrition Formula: Effect on Preoperative Weight Loss and Postoperative Pain, Complications and Analytical Acute Phase Reactants After Laparoscopic Sleeve Gastrectomy. Obes Surg. 2016 Jun;26(6):1221-7. doi: 10.1007/s11695-015-1880-7. PMID 26358120